CLINICAL TRIAL: NCT04730674
Title: Predictive Factors Affecting the Efficacy of Local Tetracycline Injection for Treatment of Post-mastectomy Seroma.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zagazig University (Other Government)
Responsible Party: Principal Investigator, Joseph Rizk Awad, lecturer of surgery, faculty of human medicine, Zagazig University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: predictors of tetracycline
Record Dates: First submitted 2021-01-16; First posted 2021-01-29 (Actual); Last update posted 2021-01-29 (Actual); Status verified 2021-01

CONDITIONS: Post-mastectomty Seroma
MeSH Terms: interventions — Lidocaine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- post-mastectomty seroma group (Experimental): female patients with established diagnosis of post-mastectomy seroma following modified radical mastectomy, were treated by local injection of tetracycline after the seroma fluid was aspirated, then a crepe bandage was applied over the mastectomy area. Then after 5 days the patient were examined again for seroma re-collection or the presence of complications. The amount of seroma aspirated in each session.
  Interventions: Drug: tetracycline mixed with xylocaine

INTERVENTIONS:
Drug: tetracycline mixed with xylocaine — 10 cc of saline containing 2 gm of tetracycline mixed with 5 ml of 2% xylocaine (as a pain relieving agent) was injected at the seroma bed.

SUMMARY:
female patients with established diagnosis of post-mastectomy seroma following modified radical mastectomy, were treated by local injection of tetracycline after the seroma fluid was aspirated, then a crepe bandage was applied over the mastectomy area. Then after 5 days the patient were examined again for seroma re-collection or the presence of complications. The amount of seroma aspirated in each session.

DETAILED DESCRIPTION:
In this study, 18 patients with established diagnosis of post-mastectomy seroma were included. All of them were females undergoing modified radical mastectomy where seroma appeared after drain removal.

The age, co-morbidities, total leukocytic count (as an indicator of infection), serum albumin and tumour size and pathology for all of them were recorded. Then we interfered with our tetracycline injection technique for the treatment of seroma.

All the patients were consented regarding this therapeutic technique explaining the expected possible occurrence of some pain during and after injection, other complications like wound infection or flap necrosis necessitating further intervention. Moreover, repetition of the technique may be needed

In our technique the following was adopted:

1. First, the seroma fluid was aspirated completely using a 20 cc syringe while the patient lying flat and the needle inserted in the most dependent area
2. Then, 10 cc of saline containing 2 gm of tetracycline mixed with 5 ml of 2% xylocaine (as a pain relieving agent) was injected at the seroma bed.
3. After completion of injection, a crepe bandage was applied over the mastectomy area (flaps covering the seroma bed)
4. Then after 5 days the patient were examined again for seroma re-collection or the presence of complications as infection or flap necrosis. If there were any re-collection, the tetracycline injection procedure would be repeated.

The amount of seroma aspirated in each session in addition to the complications if present were recorded.

ELIGIBILITY:
Inclusion Criteria:

* any patient with post-mastectomy seroma following modified radical mastectomy after removal of drain
* no signs of infection or flap necrosis

Exclusion Criteria:

* patients with post-mastectomy seroma following modified radical mastectomy with drain still in
* if signs of infection or flap necrosis present

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
The number of injection sessions to reach complete resolution of seroma | 5 days
  number of injection sessions to reach complete resolution of seroma

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine, Zagazig, Sharqia Province, Egypt

IPD SHARING:
Plan to Share IPD: Undecided